CLINICAL TRIAL: NCT00746746
Title: A Phase II Study of an Anti-Tumor Immunotherapy Regimen Comprised of Pegylated Interferon-Alpha 2b (PEG-Intron)and HyperAcute Melanoma Vaccine for Subjects With Advanced Melanoma
Brief Title: A Phase II Study of an Anti-Tumor Immunotherapy Regimen Comprised of Pegylated Interferon-Alpha 2b and HyperAcute Melanoma Vaccine for Subjects With Advanced Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ochsner Health System (Other)
Collaborators: NewLink Genetics Corporation (Industry)
Responsible Party: Adam I. Riker, M.D. Medical Director of Cancer Services, Ochsner Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USA-MCI-01; IND# 13647
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2008-09

CONDITIONS: Melanoma
Keywords: Advanced Melanoma
MeSH Terms: conditions — Melanoma | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: HyperAcute vaccine — 1.8 mL weekly
Drug: Pegylated Interferon-Alpha 2b — 6.0 mcg/kg weekly
  Other Names: PEG-Intron

SUMMARY:
The purpose of this study is to determine the safety of giving subjects with advanced, recurrent or refractory melanoma the HyperAcute® Melanoma vaccine with a variant of a drug, called Interferon (PEG-Intron®) that is specially formulated to be given on a weekly basis (instead of daily). The study vaccine (HyperAcute®-Melanoma) is made from three types of human melanoma cell lines (grown in the laboratory) in which the genes have been slightly changed. This clinical study will try to discover the safety of the study vaccine combined with PEG-Intron®, its side effects and the potential benefits, if any.

DETAILED DESCRIPTION:
This study will look at the anti-tumor vaccine effect, side effects and toxicity of the HyperAcute® Vaccine with PEG-Intron®. It is hoped that the immune system's response to these genetically engineered melanoma cells and PEG-Intron® will cause a reaction that will make it react to and attack and kill the melanoma cells and keep it from growing, possibly causing the tumors to shrink.

Patients that are eligible are 19 years or older and have been diagnosed with advanced, treatment resistant or recurrent melanoma, an aggressive usually pigmented form of skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* Histological diagnosis of melanoma
* AJCC Stage IIIC (any T, N1b, N2b, N3, M0) or Stage IV (any T, and N, M1), metastatic, progressive, refractory, recurrent or high risk of recurrence melanoma.
* Expected survival of more than 6 months
* Adequate organ function
* Measurable or non-measurable disease
* Must have negative serologies for Hepatitis B and C and HIV prior to entering study
* Must be more than 4 weeks since major surgery, radiotherapy, chemotherapy or biotherapy/targeted therapies
* Male and female subjects of child producing potential must agree to use contraception or avoidance pregnancy measures while enrolled on the study and for one month after the last immunization.

Exclusion Criteria:

* Active CNS metastases or carcinomatous meningitis
* Hypercalcemia
* Pregnant or nursing women
* Other malignancy within five years
* History of organ transplant or current active immunosuppressive therapy
* Subjects taking systemic corticosteroid therapy
* Active infection or antibiotics within 1-week prior to study
* Uncontrolled or significant congestive heart failure, myocardial infarction, ventricular arrhythmias or pulmonary dysfunction
* Autoimmune disease
* A known allergy to any component of the HyperAcute vaccine or PEG-Intron
* Patients having undergone splenectomy
* Patients with sickle-cell anemia or thalassemia major.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
To conduct scientific studies of patient tumor and peripheral blood samples to determine the mechanism of any observed anti-tumor effect involving the immune responses to the HyperAcute® vaccine alone & combined with PEG-Intron | 2 years

SECONDARY OUTCOMES:
To determine the safety and response rate of the administration of the HyperAcute®-Melanoma Vaccine combined with PEG-Intron® into patients with recurrent, refractory, metastatic, or high risk of recurrence melanoma | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Adam I Riker, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Health System, New Orleans, Louisiana, United States

REFERENCES:
- See also: Ochsner Health System website — http://www.ochsner.org